CLINICAL TRIAL: NCT05261815
Title: Comparative Effectivness Between Ultrasound Therapy And High Intensity Laser Therapy In The Treatment Of Lumbar Disc Herniation.
Brief Title: Compare Effects of Ultrasound Therapy With High Intensity Laser Therapy for Treatment of Lumbar Disc Herniation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC-FSD-00244
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Disk Herniated Lumbar
Keywords: High Intensity Laser Therapy; Ultrasound Therapy; Lumbar; Disc Herniation.; Randomized Control Trial; Comparison
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study would be double blinded as participants and assessors of the study would be kept blind of the treatment group to which the participant will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound therapy (Experimental): * Continuous ultrasound therapy for 15 minutes
  * Traction for 30 minutes
  * Spinal decompression exercises for 20 min
  Interventions: Other: Ultrasound Therapy
- High Intensity Laser Therapy (Experimental): * High intensity laser for 10 minutes
  * Traction for 30 minutes
  * Spinal decompression exercises for 20 min
  Interventions: Other: High Intensity Laser Therapy

INTERVENTIONS:
Other: Ultrasound Therapy — Ultrasound Therapy improves the pain management in patients with herniation. It eases down the severity of symptoms as well.
  Arms: Ultrasound therapy
Other: High Intensity Laser Therapy — Treatment of low disc herniation should be non-surgical, pharmacological and by physical therapy modalities. Laser radiation with high intensity used as a modality called high intensity laser therapy. It is used to relieve the pain by three process; Photo-chemical, Photo-thermal, Photo-mechanical. High Intensity Laser Therapy uses high intensity laser irradiation and low light absorption.
  Arms: High Intensity Laser Therapy

SUMMARY:
The aim of this study is to assess and compare the effects of ultrasound therapy and High Intensity Laser Therapy, as the treatment option in case of lumbar disc herniation.

DETAILED DESCRIPTION:
A randomized control trail will be conducted in Safi teaching hospital near Riphah international university, after approval of synopsis. To evaluate the comparison and effect of Ultrasound therapy and High Intensity Laser Therapy, 30 patients will be randomly assigned to High Intensity Laser Therapy and Ultrasound group. Patients will be selected according to predefined inclusion and exclusion criteria. All the patients will be evaluated by computed tomography scan or magnetic resonance of lumbar spine. Non-probability convenient sampling will be used to approach the patients in hospital. Participants received 15 treatment session of High Intensity Laser Therapy and Ultrasound therapy over a period of three consecutive weeks (five days/week). Two types of tools will be used to evaluate the find out the comparison of both groups Visual analog scale and Oswestry lowback pain disability questionnaire. Data will be collected pre-treatment and post-treatment after 15 days. Data will be analyzed by Statistical Package of Social Sciences Version 20. Difference between pre-treatment to post treatment between group will be analyzed by Mann-Whitney test, and Within group difference will be analyzed by Wilcoxon signed- rank test. The level of statistical significance will be set as p< 0.05

ELIGIBILITY:
Inclusion Criteria:

* Patient above age 18 and adult
* Patient with lumbar disc herniation diagnosed by MRI
* Patient with no history of trauma and congenital abnormalities

Exclusion Criteria:

* If patient received anesthesia or corticosteroid within 4 week
* Patient with osteoporosis
* Patient with surgery or previous fracture of spinal stenosis
* A history of acute trauma like osteoarthritis, myofascial pain syndrome, inflammatory rheumatic disease, systemic lupus erythematosus, diabetes mellitus type 1 and 2, thyroid dysfunction, obesity, pacemaker, neurological pathologies and anxious- depressive syndrome.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12th Week
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Oswestry low back pain questionnaire | 12th Week
  The Oswestry Low Back Pain Disability Questionnaire is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No